CLINICAL TRIAL: NCT07288255
Title: Application of 'One-stop' Single-lumen Endotracheal Intubation for Electromagnetic Navigation Bronchoscopy-guided Localization and Resection of Pulmonary Nodules: a Single-center Retrospective Cohort Analysis
Brief Title: Single-lumen Endotracheal Intubation in ENB-guided Localization and Resection of Pulmonary Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Ruijin Hospital, Department of Thoracic Surgery, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH-TS-202501
Record Dates: First submitted 2025-09-28; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lung Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SL-DL group (Sham Comparator): After the ENB-guided localization procedure, patients in the single-lumen to double-lumen (SL-DL) group had their single-lumen endotracheal tubes were replaced with double-lumen tubes, enabling thoracoscopic surgery to be performed in the lateral decubitus position under one-lung ventilation (OLV).
  Interventions: Procedure: single-lumen to double-lumen
- SL group (Active Comparator): The patients in the single-lumen (SL) group did not undergo tube replacement. Throughout the surgery, anesthesiologists adjusted the tidal volume to optimize the surgical field for the thoracic surgeons.
  Interventions: Procedure: Single lumen

INTERVENTIONS:
Procedure: Single lumen — patients in the single-lumen (SL) group did not undergo tube replacement. Throughout the surgery, anesthesiologists adjusted the tidal volume to optimize the surgical field for the thoracic surgeons
  Arms: SL group
Procedure: single-lumen to double-lumen — patients in the single-lumen to double-lumen (SL-DL) group had their single-lumen endotracheal tubes were replaced with double-lumen tubes, enabling thoracoscopic surgery to be performed in the lateral decubitus position under one-lung ventilation (OLV).
  Arms: SL-DL group

SUMMARY:
The goal of this clinical study is to evaluate the practicality, safety, and feasibility of a 'one-stop' single-lumen (SL) endotracheal intubation strategy for patients undergoing wedge resection of early-stage lung nodules with electromagnetic navigation bronchoscopy (ENB)-guided localization. The main question it aims to answer is:

• Is the 'one-stop' SL strategy, where an SL tube is used continuously from ENB localization through surgery, non-inferior to the conventional practice of switching from an SL to a double-lumen (DL) tube in terms of perioperative outcomes and complication rates?

Participants scheduled for ENB-guided localization followed by wedge resection will be managed with either the proposed 'one-stop' SL intubation method or the conventional SL-to-DL conversion method. Researchers will compare key perioperative indicators and patient outcomes between the two groups.

DETAILED DESCRIPTION:
With increased health awareness and the widespread use of low-dose CT for lung cancer screening, early detection rates have risen. For early-stage non-small cell lung cancer, sub-lobar resection (segmentectomy or wedge resection) is now strongly recommended for peripheral nodules ≤2 cm without nodal involvement, as per recent landmark trials and NCCN guidelines. However, for wedge resection, precise localization and minimization of pulmonary function impairment still pose challenges for thoracic surgeons. Therefore, achieving effective resection while preserving lung function as much as possible necessitates precise localization of pulmonary nodules.

The CT-guided hook-wire localization method is currently the most frequently used technique in clinical practice for pulmonary nodule localization, but patients may experience significant pain and there is a risk of dislodgement of the hook wire during patient transfer or positioning before surgery. Furthermore, CT localization results in a high risk of pneumothorax and bleeding. The emergence of electromagnetic navigation bronchoscopy (ENB) not only alleviates patient discomfort but also reduces surgical time and lowers the risk of complications.

Typically, during ENB-guided localization, a single-lumen (SL) endotracheal tube is used under general anesthesia and subsequently replaced with a double-lumen (DL) endotracheal tube after the procedure. However, the conversion from SL to DL could potentially elevate the possibility of airway damage and anesthetic complications. Therefore, in patients undergoing wedge resection with ENB-guided localization, the investigators propose a 'one-stop' SL strategy, in which an SL tube is employed throughout the entire process from localization to surgery.

This study aimed to evaluate the practicality of utilizing SL endotracheal intubation for the entire process of ENB-guided localization and subsequent surgical procedure, referred as 'one-stop' SL. By comparing the conventional practice of the transition from SL to DL intubation with our proposed 'one-stop' SL intubation method based on perioperative indicators and patient outcomes, the investigators hope to determine whether the 'one-stop' SL strategy is safe and feasible clinically.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had pulmonary nodules and underwent video-assisted thoracoscopic surgery (VATS) lung surgery with ENB-guided nodule localization

Exclusion Criteria:

* Patients who received non-intubated anesthesia or underwent wedge resection combined with lobectomy or segmentectomy were excluded.
* Perioperative data were missing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative complications | Within 30 days postoperatively
  Postoperative complications included the incidence of complications such as pneumonia, atelectasis, pneumothorax, air leakage, and pleural effusion.

SECONDARY OUTCOMES:
Pain score | Perioperative
  Pain score was assessed using the Visual Analog Scale (VAS), a 10-point scale where 0 represents "no pain" and 10 represents "the worst pain imaginable," with higher scores indicating more severe pain.
Semiquantitative cough strength score | Perioperative
  Cough strength was evaluated using the semiquantitative cough strength score (SCSS), graded from 0 (weak) to 5 (strong)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: With publication
Access Criteria: Interested investigators will be required to submit a formal letter of intent outlining research aims, rationale, and approach. Furthermore, documentation of local IRB approval, including a description of type of review, should be submitted with the data request.